CLINICAL TRIAL: NCT00764751
Title: LEO 19123 Cream in the Treatment of Psoriasis Vulgaris
Brief Title: Efficacy and Safety of LEO 19123 Cream in the Treatment of Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEO 19123-C24
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: LEO 19123 Cream (calcipotriol plus LEO 80122)
- 2 (Active Comparator)
  Interventions: Drug: Dovonex® cream
- 3 (Placebo Comparator)
  Interventions: Drug: Cream vehicle

INTERVENTIONS:
Drug: LEO 19123 Cream (calcipotriol plus LEO 80122) — Once daily application
  Arms: 1
Drug: Dovonex® cream — Twice daily application
  Arms: 2
Drug: Cream vehicle — Twice daily application
  Arms: 3

SUMMARY:
This study will compare the efficacy and safety of once daily treatment of LEO 19123 cream versus Dovonex® cream (applied twice daily) and versus LEO 19123 cream vehicle alone (applied twice daily) in subjects with psoriasis vulgaris. Subject will be treated for 4 weeks. All subjects will apply LEO 19123 cream to psoriasis lesions on the left or right side of the body and either Dovonex® cream or cream vehicle to lesions on the other side.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent to be obtained prior to any trial related procedure, including washout.
* Clinical diagnosis of psoriasis vulgaris involving trunk and/or arms and/or legs with a symmetrical distribution amenable to treatment with a maximum of 50 g/week of topical medication on each side of the body. At Visit 1, there should not be a difference between the right and left side of more than 1 for each of the PASI criteria (redness, thickness and scaliness).
* A minimum PASI score for extent of 2 on each side in at least one body region (i.e. psoriasis affecting at least 10% of left and right arm, and/or 10% of left and right side of the trunk, and/or 10% of left and right leg).
* Disease severity graded mild, moderate, severe or very severe according to the Investigator's global assessment (IGA) of disease severity on each side of the body. The assessment should be the same for both sides of the body.
* Age 18 years or above
* Male subjects, or females of non-childbearing potential (i.e. surgically sterile or at least two years postmenopausal)
* Attending a hospital outpatient clinic or the private practice of a dermatologist

Exclusion Criteria:

* Subjects using systemic treatments with biological therapies with a possible effect on psoriasis vulgaris within 12 weeks prior to randomisation (e.g. alefacept, efalizumab, etanercept, infliximab, adalimumab)
* Systemic treatment with all other therapies, besides biologics, with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within 4 weeks prior to randomisation (inhaled or intranasal steroids for asthma or rhinitis may be used)
* PUVA or Grenz ray therapy within 4 weeks prior to randomisation
* UVB therapy within 2 weeks prior to randomisation
* Any topical treatment (except for emollients) of the trunk/limbs (except on flexures) within 2 weeks prior to randomisation
* Topical treatment for other relevant skin disorders on the face and flexures (e.g., facial and flexural psoriasis, eczema) with potent or very potent (WHO group III-IV) corticosteroids, vitamin D analogues or retinoids within 2 weeks prior to randomisation
* Topical treatment for other relevant skin disorders on the scalp (e.g. scalp psoriasis) with very potent (WHO group IV) corticosteroids, vitamin D analogues or retinoids within 2 weeks prior to randomisation
* Planned initiation of, or changes to concomitant medication that could affect psoriasis vulgaris (e.g., beta blockers, ACE inhibitors, anti-malaria drugs, lithium) within 2 weeks prior to randomisation
* Subjects who have received treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within the 4-week period prior to randomisation
* Subjects with current participation in any other interventional clinical trial
* Subjects with any of the following conditions present on the treatment area: eczematous skin, atopic dermatitis, clinical infection, ulcers and wounds
* Subjects with a history of serious allergy, allergic skin rash or sensitivity to any component of the investigational products or formulations being tested
* Subjects with positive hepatitis B, C or HIV
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia
* Current diagnosis of erythrodermic, exfoliative, guttate or pustular psoriasis
* Planned exposure to the sun during the study that may affect psoriasis vulgaris (i.e., normal lifestyle outdoor activities are permitted but deliberate exposure to sunlight or artificial ultraviolet light should be avoided)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodion Kunynetz, MD, Principal Investigator — UltraNova Skincare
Locations (1):
- UltraNova Skincare, Barrie, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: * LEO 19123 (calcipotriol 50 mcg/g plus LEO 80122 0.6 mg/g) cream for topical application once daily in the evening to lesions on one side of the body. Maximum 50 g/week
  * Dovonex® (calcipotriol 50 mcg/g) cream for topical application twice daily to the lesions on the other side of the body. Maximum 50 g/week.
- Group B: * LEO 19123 (calcipotriol 50 mcg/g plus LEO 80122 0.6 mg/g) cream for topical application once daily in the evening to lesions on one side of the body. Maximum 50 g/week.
  * LEO 19123 cream vehicle for topical application twice daily to the lesions on the other side of the body. Maximum 50 g/week.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 39 | 12
Completed | 37 | 11
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Psoriasis flare up on the scalp | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 39 | 12 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (14.3) | 57.7 (9.8) | 54.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 28 | 9 | 37
Region of Enrollment [Number; unit: participants]
  Canada | 39 | 12 | 51

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change in PASI (Psoriasis Area Severity Index)
Description: The following formula was used to calculate the PASI for each side of the body:
  Upper extremities: 0.2 (R + T+ S) E = X Trunk: 0.3 (R + T+ S) E = Y Lower extremities 0.4 (R + T+ S) E = Z
  where: R = score for redness T = score for thickness S = score for scaliness E = score for extent
  The sum of X + Y + Z gives the total PASI, which can range from 0 to 64.8. The PASI used in this study is modified to exclude assessment of the head, as study treatment was not used here.
Time Frame: From baseline (Day 0) to end of treatment (Day 28)
Measure: Mean (Standard Deviation); unit: percentage change in PASI
Groups:
- Group A: LEO 19123; Group B: LEO 19123: LEO 19123 (calcipotriol 50 mcg/g plus LEO 80122 0.6 mg/g) cream for topical application once daily in the evening to lesions on one side of the body. Maximum 50 g/week
- Group A: Dovonex®: Dovonex® (calcipotriol 50 mcg/g) cream for topical application twice daily to the lesions on the other side of the body. Maximum 50 g/week.
- Group B: LEO 19123 Vehicle: LEO 19123 cream vehicle for topical application twice daily to the lesions on the other side of the body. Maximum 50 g/week.
Arm/Group | Group A: LEO 19123 | Group A: Dovonex® | Group B: LEO 19123 | Group B: LEO 19123 Vehicle
Number analyzed (Participants) | 39 | 39 | 12 | 12
percentage change in PASI | -24.8 (33.2) | -40.2 (27.8) | -46.8 (27.0) | -29.8 (20.9)
Statistical Analysis 1: Comparison: Group A: LEO 19123 vs Group A: Dovonex®; Test type: Superiority; p = 0.003, Paired t-test; Mean Difference (Final Values) = 15.4, 95% CI 2-sided [5.6 to 25]
Statistical Analysis 2: Comparison: Group B: LEO 19123 vs Group B: LEO 19123 Vehicle; Test type: Superiority; p = 0.07, Paired t-test; Mean Difference (Final Values) = -17.1, 95% CI 2-sided [-36.0 to 1.9]

2. Secondary Outcome: Investigator's Global Assessment of Disease Severity
Description: At all visits the (sub)investigator made a global assessment of the disease severity for psoriasis on the left and right side, respectively, of the body by use of the 6-point scale below. These assessments were to represent the average lesion severity on the left and right side, respectively. These assessments were to be based on the condition of the disease at the time of evaluation, and not in relation to the condition at a previous visit.
  Clear Almost clear Mild Moderate Severe Very severe
Time Frame: At end of treatment (Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: LEO 19123 | Group A: Dovonex® | Group B: LEO 19123 | Group B: LEO 19123 Vehicle
Number analyzed (Participants) | 39 | 39 | 12 | 12
Participants
  Clear | 0 | 0 | 0 | 0
  Almost clear | 3 | 1 | 4 | 0
  Mild | 8 | 17 | 3 | 5
  Moderate | 24 | 20 | 5 | 5
  Severe | 4 | 1 | 0 | 2
  Very severe | 0 | 0 | 0 | 0

3. Secondary Outcome: Participants With "Controlled Disease" According to the Investigator's Global Assessment of Disease Severity
Description: For subjects with a baseline (Visit 1) severity of moderate or worse, "controlled disease" is defined as "clear" or "almost clear" according to the Investigator's global assessment of disease severity. For subjects with a baseline (Visit 1) severity of mild, "controlled disease" is defined as "clear" according to the Investigator's global assessment of disease severity.
Time Frame: At end of treatment (Day 28)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: LEO 19123 | Group A: Dovonex® | Group B: LEO 19123 | Group B: LEO 19123 Vehicle
Number analyzed (Participants) | 39 | 39 | 12 | 12
Participants
  Controlled disease | 2 | 1 | 4 | 0
  No controlled disease | 37 | 38 | 8 | 12

4. Secondary Outcome: Participant's Overall Assessment of Treatment Response
Description: The participant assessed the treatment response by use of the 6-point scale below.
  Worse Unchanged Slight improvement Moderate improvement Marked improvement Almost clear Cleared
Time Frame: At end of treatment (Day 28)
Population: All randomized participants have been included in the analysis. One participant withdrew and did therefore not give their assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: LEO 19123 | Group A: Dovonex® | Group B: LEO 19123 | Group B: LEO 19123 Vehicle
Number analyzed (Participants) | 39 | 39 | 12 | 12
Participants
  Worse | 2 | 1 | 1 | 0
  Unchanged | 9 | 4 | 3 | 3
  Slight improvement | 12 | 9 | 1 | 7
  Moderate improvement | 12 | 12 | 5 | 1
  Marked improvement | 3 | 12 | 2 | 1
  Almost clear | 0 | 0 | 0 | 0
  Clear | 0 | 0 | 0 | 0

5. Secondary Outcome: Participant's Assessment of Treatment Preference
Time Frame: At end of treatment (Day 28)
Population: All randomized participants have been included in the analysis. One participant withdrew and did therefore not give their preference.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 39 | 12
Participants
  LEO 19123 | 5 | 6
  No preference | 12 | 3
  Reference product | 21 | 3

6. Secondary Outcome: Participants With at Least 75% Reduction in PASI (PASI 75)
Time Frame: From baseline (Day 0) to end of treatment (Day 28)
Population: Two participants withdrew from the LEO 19123 versus Dovonex® group at Week 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: LEO 19123 | Group A: Dovonex® | Group B: LEO 19123 | Group B: LEO 19123 Vehicle
Number analyzed (Participants) | 39 | 39 | 12 | 12
Participants
  >=75% PASI reduction | 2 | 4 | 1 | 0
  75% PASI reduction | 37 | 35 | 11 | 12

7. Secondary Outcome: Participants With at Least 50% Reduction in PASI (PASI 50)
Time Frame: From baseline (Day 0) to end of treatment (day 28)
Population: All randomised participants have been included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: LEO 19123 | Group A: Dovonex® | Group B: LEO 19123 | Group B: LEO 19123 Vehicle
Number analyzed (Participants) | 39 | 39 | 12 | 12
Participants
  >= 50% PASI reduction | 9 | 15 | 7 | 2
  < 50% PASI reduction | 30 | 24 | 5 | 10

8. Secondary Outcome: The Absolute Change in PASI (Psoriasis Area Severity Index)
Description: as for outcome 1
Time Frame: From baseline to end of treatment (Day 28)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: LEO 19123 | Group A: Dovonex® | Group B: LEO 19123 | Group B: LEO 19123 Vehicle
Number analyzed (Participants) | 39 | 39 | 12 | 12
units on a scale | -2.6 (4.0) | -3.8 (3.6) | -4.2 (2.9) | -2.5 (2.1)

ADVERSE EVENTS:
Time Frame: From Day 0 to follow up (Day 28+14)
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/12
Other Adverse Events (participants affected / at risk) | 15/38 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=38) | Group B (N=12)
Cholecystitis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=38) | Group B (N=12)
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submit-ted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.